CLINICAL TRIAL: NCT02890615
Title: Effectiveness of a Telephone-supported Depression Self-care Intervention for Cancer Survivors
Brief Title: CanDirect: Effectiveness of a Telephone-supported Depression Self-care Intervention for Cancer Survivors
Acronym: CanDirect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Jane McCusker, MD DrPH, Professor Emerita and Full Professor Post-Retirement, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SMHC 16-15
Record Dates: First submitted 2016-08-24; First posted 2016-09-07 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Depression
Keywords: Survivors; Self Care
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Depression Self-care Intervention (SCI) (Experimental): Intervention group participants will receive the Depression Self-Care Toolkit for Cancer Survivors and will be supported by telephone by a coach who will help to activate them, guide them through the materials, help in selecting appropriate tools, and provide positive reinforcement. Coach contacts will be made every week for 3 months followed by 3 monthly contacts, up to a maximum of 15 contacts, lasting 10-20 minutes each.
  The coach uses a stepped approach (i.e. educate about depression, initiate mood monitoring, determine participant's goals with respect to reducing depressive symptoms, and help with the use of specific tools). A suggested script is provided for the coach as a framework for each call. Tailoring of the SCI to different participants will be based on problems, depressive symptoms (from the PHQ-9), or concerns a participant may raise during the call.
  Interventions: Behavioral: Depression self-care
- Control group (No Intervention): Members of both groups will continue to receive "usual care" for their depression. We will not interfere with usual care beyond recommending that participants discuss their depressive symptoms with their doctor. If participants consent, a short progress report will be send to their treating physician at the end of the study. At each follow-up, we will ask participants about specific treatment they have received for depression since entering the study (antidepressant medication initiation, discontinuation, change of dose, or psychotherapy) and use of community resources. The Intervention group will receive the Depression SCI. The Control group will receive only usual care for 6 months after randomization; they will be given the Toolkit with a single coaching call upon completion of the final interview, to ensure their access to depression treatment.

INTERVENTIONS:
Behavioral: Depression self-care — Toolkit and coaching
  Arms: Depression Self-care Intervention (SCI)

SUMMARY:
Depressive symptoms are common in cancer survivors; 15% or more of cancer patients, even 1 year after diagnosis, experience depressive symptoms that can have a negative impact on their quality of life. Canadian care guidelines for cancer survivors recommend supporting the active engagement of survivors in their self-care.

This study is an evaluation of the effect of a depression self-care program which includes a self-care toolkit and support in the form of regular telephone calls from a self-care coach.

The toolkit contains tools that help cancer survivors:

1. Learn new information to better understand depression. This can help people feel that they are not alone, and that their experience is not abnormal. Better understanding a condition also helps people feel more confident in their communications with health care professionals and can make it easier to share their experience with family and friends.
2. Learn and practice new coping skills. This can help people feel confident that they can engage in the behaviours that have been shown to be beneficial for mood, e.g. restructuring thoughts, problem solving, and planning pleasant activities.

People eligible for the study are aged 18 and over, 1-10 years post-diagnosis, have completed primary cancer treatment (chemotherapy, radiation therapy or surgery) for any type of cancer, and have moderate depressive symptoms (as measured by a Patient Health Questionnaire (PHQ-9) score of 8-19). Recruitment will be conducted at cancer care centres in Montreal and at the Princess Margaret Cancer Centre in Toronto, and via community cancer support groups in Quebec and Ontario. Each participant enrolled in the study will receive the self-care toolkit (half will receive the toolkit and support calls at the start of the study, and half will receive the toolkit at the end), and will be followed for 6 months.

This proposed self-care program is innovative in its approach to the treatment of depression and has the potential to significantly improve the quality of life for Canadian cancer survivors with persistent depressive symptoms. The results of the study will determine whether the supported depression self-care program for cancer survivors is effective. The program is designed to be sustainable and widely applicable as it involves minimal costs, and the coaching can be delivered by telephone by volunteers in hospital and community settings. Investigators will work with clinical stakeholders and patient representatives to ensure that deliverables are relevant to the target population. Specific deliverables (in both French and English) include: a toolkit with a manual describing its use; a manual detailing coaching procedures; reports for decision makers and community cancer care groups; and short summaries for stakeholder groups.

DETAILED DESCRIPTION:
This pragmatic randomized controlled superiority trial aims to assess the effectiveness of a telephone-supported depression SCI in cancer survivors with moderate depressive symptoms when given in addition to usual care, in comparison to usual care only. Because of the pragmatic nature of this trial, members of both groups will continue to receive "usual care" for their depression, which may vary widely depending on local resources and medical practice. At each follow-up, participants are asked about specific treatment they have received for depression since entering the study (antidepressant medication initiation, discontinuation, change of dose, or psychotherapy) and their participation in community support groups and related activities; investigators will explore whether this care mediates the effects of the intervention. The study includes safeguards for participants who become suicidal or severely depressed during the study.

Research questions

Among cancer survivors in the post-treatment phase who have moderate to moderately-severe depressive symptoms [Patient Health Questionnaire (PHQ-9) score 8-19]:

1. Primary research question: What is the effect of a telephone-supported depression self-care intervention (SCI) plus usual care compared to usual care only (control group CTL) on the primary outcome - severity of depression symptoms as measured by the Centre for Epidemiologic Studies Depression Scale (CES-D) 6 months after randomization? Hypothesis: Participants who receive the SCI will have better 6 month primary outcomes than those randomized to the Control group.
2. Secondary questions:

   1. What are the effects of the SCI on: CES-D score at 3 months; depression diagnosis at 6 months; and mental health related quality of life, activation, severity of anxiety symptoms at 3 and 6 months, and use of health services over 6 months? Hypothesis: Participants who receive the SCI will have better health outcomes and lower use of health services than those randomized to the Control group.
   2. Are the effects of the SCI on the primary outcome modified by 5 primary baseline patient characteristics [major depression diagnosis; antidepressant medication; activation; recruitment source (clinical vs community); and level of education ] or by 9 secondary patient characteristics [cancer type, ongoing adjuvant cancer treatment (yes, no), years from cancer diagnosis (quartiles), severity of anxiety (as measured by the Hospital Anxiety and Depression Scale - Anxiety subscale (HADS-A)), physical health-related quality of life (as measured by the Physical Component Summary (PCS) of the Short Form Health Survey (SF-12)) (quartiles), sex, age (quartiles), family support for self-management (quartiles), province of residence (Quebec, Ontario)].

      Hypothesis and support Effect moderators (or modifiers) represent variables e.g. patient characteristics, measured at baseline, that interact with treatment to change outcome for each sub-group. These specify for whom treatment is most effective and can improve power in subsequent trials by better selection of study groups for stratification. In selecting those potential modifiers/moderators that will be pre-specified for testing, investigators followed consensus criteria for assessment of these factors. Pinctus proposes 5 criteria for systematic reviews of randomized controlled trials confirming moderator effects: 1) was the analysis a priori; 2) was selection of factors for analysis clinically plausible and either theory-based or evidence-based; 3) were moderators measured prior to randomization; 4) adequate quality of measurement; 5) explicit test of the interaction between moderator and treatment. For meta-analyses exploring moderator effects, criteria 1 and 2 are not required.

      Investigators will analyze 5 possible moderators using sub-group analyses:

      Major depression They hypothesize that the intervention will be more effective among participants with a diagnosis of major depression (measured through the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders Disorders - Major Depressive Syndrome in the Mood Disorders Module (SCID)) than those without. A meta-analysis of psychosocial interventions in cancer populations found that studies in which patients were pre-selected for higher levels of distress found greater effectiveness of the intervention. A meta-analysis of depression self-care interventions also reported greater effectiveness in patients with major depression, although only in univariate analysis.

      Antidepressant medication Investigators hypothesize that the intervention will be more effective among participants with baseline antidepressant medication than those without. A meta-analysis found that the combination of psychotherapy and pharmacotherapy is more effective in the treatment of depression than psychotherapy alone.

      Activation Investigators hypothesize that the intervention will be more effective among participants with higher baseline activation than those with lower levels. As there is no accepted cut-point on the Patient Activation Measure (PAM) scale, higher activation will be defined as a PAM score in the highest quartile. In a randomized controlled trial of the depression self-care intervention among primary care patients with chronic physical conditions, investigators found that coaching was more effective among patients with higher baseline self-efficacy (one component of activation).

      Recruitment source Investigators hypothesize that the intervention will be more effective among participants recruited from community settings than from clinical settings. A meta-analysis of depression self-care interventions also reported lower effectiveness in patients studied in clinical settings, although only in univariate analysis. Participants recruited from community settings in this study (e.g., from community groups and social media) will already be selected to be more motivated to participate actively in the intervention.

      Level of education Investigators hypothesize that the intervention will be more effective among participants with higher education, defined as some education beyond high school (e.g, diploma or university), compared with those with only high school or less education. Investigators are not aware of evidence supporting this hypothesis, but the use of paper and pencil and electronic tools will be more familiar to those with a higher level of education.

      In addition to these 5 hypothesized moderators, investigators propose to examine the following 9 secondary potential baseline moderators, each with a maximum of 4 categories:

      cancer type, ongoing adjuvant cancer treatment (yes, no), years from cancer diagnosis (quartiles), severity of anxiety (HADS), physical health-related quality of life (PCS) (quartiles), sex, age (quartiles), family support for self-management (quartiles), province of residence (Quebec, Ontario).
   3. In the Intervention group, is greater adherence to the SCI (e.g., use of self-care tools, completion of written exercises and mood monitoring, goal setting, greater number of coaching contacts) associated with better primary and secondary outcomes? Hypothesis: Participants who adhere to the SCI, particularly those who actively engage with the Cognitive behavioural therapy (CBT)-based tools will have greater reductions in depressive symptoms, diagnoses, and severity of anxiety symptoms, and greater increases in activation and quality of life.
3. Economic analysis:

An economic analysis of the SCI is beyond the scope of this study. In the current study, investigators collect patient-reported data on use of health services and request additional (optional) consent for linkage to health care administrative data (the Ontario Health Insurance Plan (OHIP) Claims database and the Discharge Abstract Database (DAD)). They plan to seek additional funding for analyses of these use of services and administrative data for a future study on impact of the SCI on use of services. They will only extract use of services data for patients who consent to this optional element, and only for a period 12 months before and 12 months after the date of enrolment in the present trial. Patients who consent to use of their administrative data are asked to provide their OHIP number to allow researchers to extract the required data.

ELIGIBILITY:
Inclusion criteria:

* completed primary cancer treatment (surgery, radiation and/or chemotherapy) for any type of cancer (NB: patients receiving adjuvant therapies will be eligible),
* between 1-10 years post-diagnosis (as suggested by clinicians collaborating on the project),
* with moderate depressive symptoms (PHQ-9 score of 8-19).

Exclusion criteria:

* metastatic disease,
* suicidal,
* moderate-severe cognitive impairment,
* unable to speak and read in English or French,
* only non-melanoma skin cancer (without any other single primary cancer),
* receiving ongoing psychological treatment at baseline (because of recent finding that this treatment may negatively modify the effectiveness of the coaching component of the intervention). NB: those who begin psychological treatment during follow-up will not be withdrawn.
* dose of antidepressant medication changed within last 6 weeks at baseline. NB: those who change dose or treatment during follow-up will not be withdrawn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2016-07; Primary Completion 2019-04 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in severity of depression symptoms: Centre for Epidemiologic Studies Depression Scale (CES-D) | Baseline, 3 months, 6 months

SECONDARY OUTCOMES:
Change in severity of anxiety symptoms: Hospital Anxiety and Depression Scale - Anxiety subscale (HADS-Anxiety) | Baseline, 3 months, 6 months
Change in mental and physical health-related quality of life: Short Form health survey (SF-12) | Baseline, 3 months, 6 months
Change in activation: Patient Activation Measure (PAM) | Baseline, 3 months, 6 months
Change in depression diagnosis: Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders - IV Disorders (SCID) | Baseline, 6 months
Change in use of health services: self-report | Baseline, 3 month, 6 month
  doctor office and clinic visits, emergency room visits, hospitalizations, psychosocial treatment or support group participation, changes in cancer diagnosis or treatment

CONTACTS AND LOCATIONS:
Locations (1):
- St Mary's Research Centre, Montreal, Quebec, Canada

REFERENCES:
- [Derived] McCusker J, Jones JM, Li M, Faria R, Yaffe MJ, Lambert SD, Ciampi A, Belzile E, de Raad M. CanDirect: Effectiveness of a Telephone-Supported Depression Self-Care Intervention for Cancer Survivors. J Clin Oncol. 2021 Apr 1;39(10):1150-1161. doi: 10.1200/JCO.20.01802. Epub 2021 Feb 8. PMID 33555912